CLINICAL TRIAL: NCT06579014
Title: Prevalence and Prognostic Effects of Thyroid Abnormalities in Patients With Acute Coronary Syndrome.
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Heba Ebraheem Badran, Principal investigator, Assiut University
Other Study IDs: Thyroid abnormalities and ACS
Record Dates: First submitted 2024-08-27; First posted 2024-08-30 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Thyroid Dysfunction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is knowledge of Prevalence of throid abnormalities in patients with acute coronary syndrome And prognostic effects of thyroid abnormalities in patients with acute coronary syndrome as early detection and management of thyroid abnormalities can improve clinical outcomes.

DETAILED DESCRIPTION:
Acute coronary syndrome (ACS) is an umbrella term used to describe a range of conditions associated with sudden, reduced blood flow to the heart. ACS includes conditions such as: Unstable Angina, Non-ST-Elevation Myocardial Infarction (NSTEMI) And ST-Elevation Myocardial Infarction (STEMI). The morbidity and mortality due to ACS are substantial-nearly half of all deaths due to coronary heart disease occur following an ACS .

Thyroid abnormalities, particularly hypothyroidism and hyperthyroidism, are relatively common in patients with ACS. Studies indicate that thyroid dysfunction can affect cardiovascular health, influencing the risk and prognosis of ACS. Reports suggest prevalence rates of Hypothyroidism 10-20% and Hyperthyroidism range from 1-5% in ACS patients .

Hypothyroidism is associated with elevated cholesterol levels, increased vascular stiffness, and heightened inflammation, can lead to reduced cardiac output and heart rate and increased incidence of heart failure and arrhythmias. all of which can exacerbate coronary artery disease and contributing to worse outcomes during ACS event. Hypothyroid patients often have a slower recovery and poorer response to standard ACS treatments, including thrombolytics and antiplatelet therapy.

Hyperthyroidism raises heart rate and contractility, leading to increased myocardial oxygen demand, which can worsen ischemia during ACS, Patients are more susceptible to arrhythmias, which can complicate ACS and lead to higher morbidity and mortality, Hyperthyroidism can cause vascular endothelial dysfunction, increasing the risk of thrombotic events during ACS and Patients may respond differently to standard ACS therapies, necessitating careful monitoring and potential adjustment of treatment strategies.

Patients with concurrent thyroid dysfunction often experience higher morbidity and mortality rates, So thyroid function should be routinely assessed in ACS patients, as early detection and management of thyroid abnormalities can improve clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ACS: (STEMI_NSTEMI)

Exclusion Criteria:

* 1-patients with cardiogenic shock. 2- patients with other endocrinal diseases. 3- patients on dialysis. 4-patients with Acute malignancy. 5-patient with thyroid diseases on treatment. 6- patients with liver diseases. 7-patients with Any autoimmune diseases

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient with ACS and thyroid abnormalities. patients with ACS and euthyroid.
Sampling Method: Non-Probability Sample
Enrollment: 129 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Prevalence of thyroid abnormalities in patients with acute coronary syndrome . | 1/9/2024-1/10/2025
  Prevalence of thyroid abnormalities in patients with acute coronary syndrome .

CONTACTS AND LOCATIONS:
Overall Officials: Rowyda Elsayed, Dr, Study Director — Assiut University